CLINICAL TRIAL: NCT03795623
Title: Voices of Patients' Relatives to Support Weaning From Mechanical Ventilation in Patients With Severe Brain Injury - VOICE-WEANING, a Randomized Clinical Trial
Brief Title: Voices of Patients' Relatives to Support Weaning From Mechanical Ventilation
Acronym: VOICE-WEANING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Hagen B. Huttner, Principal Investigator, University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 417_18 B
Record Dates: First submitted 2018-12-31; First posted 2019-01-08 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Ventilator Weaning; Weaning Failure; Brain Injuries
Keywords: Critical Illness; Respiration Disorder; Neurology
MeSH Terms: conditions — Brain Injuries; Critical Illness; Respiration Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional arm (Sham Comparator): Muted audio recordings of the patients relatives.
  Interventions: Other: Sham control
- Voice-Weaning arm (Experimental): Audio recordings of the patients relatives including information on the patient's condition and recurrent request to breath in and out.
  Interventions: Other: Voice-Weaning

INTERVENTIONS:
Other: Voice-Weaning — Audio recordings of patients' relatives for 10 minutes x 3 daily from initiation of assisted mechanical ventilation to extubation or ICU discharge.
  Arms: Voice-Weaning arm
Other: Sham control — Muted audio recordings of patients' relatives for 10 minutes x 3 daily from initiation of assisted mechanical ventilation to extubation or ICU discharge.
  Arms: Conventional arm

SUMMARY:
Patients with severe brain injuries, such as ischemic stroke and intracranial hemorrhage, frequently require mechanical ventilation. Weaning of stroke patients is complicated by impaired consciousness and respiratory drive. Higher rates of weaning failure and delayed extubation (≥ 48h) lead to ventilator associated pneumonia, higher mortality and necessity of tracheostomy.

Therefore, improving the weaning of stroke patients from mechanical ventilation is warranted to prevent ventilator-associated complications and eventually improve clinical outcomes.

This single-center, randomized, clinical trial aims at demonstrating that voices of patients' relatives support weaning from mechanical ventilation and reduce weaning failure in brain-injured patients.

DETAILED DESCRIPTION:
Methods: Adult ICU-patients with controlled mechanical ventilation ≥48h due to a neurological disease will be included in the intensive care unit. A predefined text - including information on the patient's condition and recurrent request to breath in and out - will be recorded as an audio file by one of the patient's relatives. Patients will be randomly assigned in a 1:1 ratio to the conventional treatment arm or the Voice-Weaning arm. In the conventional arm, audio recordings will be muted by an independent person resulting in a mute recording without audio signals.

When conversion from controlled to assisted mechanical ventilation is intended according to standard treatment, audio recordings will be administered in repeat mode for 10 minutes and performed three times per day. If spontaneous breathing trials (SBT) are intended according to standard treatment, the audio recordings will be played during the SBT three times per day.

Criteria for weaning not to be intended - according to Boles et al. (Weaning from mechanical ventilation. Eur Respir J. 2007) and adapted to neurological patients:

Objective measurements:

* Unstable clinical condition

  * Cardiovascular status (fC≥140/min, systolic BP <90mmHg or >180mmHg, more than minimal vasopressors)
  * Metabolic status (e.g. inacceptable electrolytes)
* Inadequate oxygenation

  * SaO2 ≤90% on FiO2 >40% or pO2/FiO2 <150mmHg or pO2/FiO2 <120mmHg in case of chronic hypoxemia (Horowitz index)
  * PEEP>8cmH2O
* Inadequate pulmonary function

  * fR ≥35/min
  * MIP>(-20 -) -25cmH2O
  * VT ≤5ml/kgKG
  * VC ≤10ml/kgKG
  * fR/VT ≥105 breaths/min x l (RSBI)
  * significant respiratory acidosis (pH≤7.25)
* Unstable neurological condition

  * sedation or inadequate mentation on sedation
  * present or anticipated intracranial mass effect (e.g. midline shift >10mm or progression, basal cistern effacement or oculomotor disturbance, signs of transfalxial/transtentorial/transforaminal herniation
  * elevation of intracranial pressure (>20 cmH2O) and/or obstructive hydrocephalus
  * severe vasospasms (>6 kHz in transcranial Doppler, or determined by CT-A/CT-P)
  * status epilepticus (determined by EEG)
  * acute intracranial infection (without established and/or treated origin)

Clinical assessment:

* Inadequate cough
* Excessive tracheobronchial secretion
* Disease acute phase for which the patient was intubated

Ethics Approval: The Institutional Review Board of the Friedrich-Alexander-Universität Erlangen-Nürnberg approved of the study on 13 November 2018.

Sample Size Calculation: The sample size is computed with 80% power and a 5% α-risk for the hypothesis of Voice Weaning achieving a 15% absolute weaning failure reduction. The sample size is increased by 10% to correct for dropouts and lost to follow up: a maximum of 354 patients will be included and an interim analysis be performed after inclusion of 50% of the calculated subjects.

ELIGIBILITY:
Inclusion Criteria:

* Intubation and controlled mechanical ventilation ≥48h due to a neurological disease
* Weaning from mechanical ventilation intended by the attending physician
* Obtained informed consent from the legal representative

Exclusion Criteria:

* Age < 18 years
* History of psychiatric disease
* Weaning from mechanical ventilation not intended or decision to limit therapeutic interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Rate of weaning failure | first 28 days after start of ventilation, or until 48 hours after extubation, or discharge from intensive care, whichever came first
  Reintubation and/or resumption of ventilatory support following extubation or death following extubation or failed spontaneous breathing trial

SECONDARY OUTCOMES:
Time of controlled ventilation | first 28 days after start of ventilation or discharge from intensive care, whichever came first
Rate of tracheotomy | first 28 days after start of ventilation or discharge from intensive care, whichever came first
  Proportion of patients requiring tracheotomy performed as percutaneous dilatative tracheotomy or surgical tracheotomy
All cause mortality rate at 90 days | first 90 days after start of ventilation
Rate of ICU delirium | first 28 days after start of ventilation or discharge from intensive care, whichever came first
  Development of delirium according to the Confusion Assessment Method for intensive care unit (CAM-ICU)

CONTACTS AND LOCATIONS:
Overall Officials: Hagen B. Huttner, MD, PhD, Principal Investigator — University of Erlangen-Nürnberg Medical School, Department of Neurology, Germany; Joji B. Kuramatsu, MD, Principal Investigator — University of Erlangen-Nürnberg Medical School, Department of Neurology, Germany; Maximilian I. Sprügel, MD, Principal Investigator — University of Erlangen-Nürnberg Medical School, Department of Neurology, Germany
Locations (1):
- University of Giessen, Giessen, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Because of local ethics committees restrictions the final decision upon release of the raw data has not been made.